CLINICAL TRIAL: NCT03730753
Title: Programmed Intermittent Epidural Bolus Versus Continuous Infusion When Added to Patient-controlled Epidural Analgesia on Bupivacaine Consumption in Labour Analgesia: a Randomized Controlled Trial
Brief Title: Programmed Intermittent Epidural Bolus Versus Continuous Infusion in Labour Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Geneviève Rivard, Principal investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018 - 2686
Record Dates: First submitted 2018-10-27; First posted 2018-11-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (Active Comparator): Continuous infusion + patient controlled epidural analgesia
  Interventions: Device: Continuous infusion
- Study group (Experimental): Programmed intermittent epidural bolus + patient controlled analgesia
  Interventions: Device: Programmed intermittent epidural bolus

INTERVENTIONS:
Device: Programmed intermittent epidural bolus — Programmed intermittent epidural bolus added to patient controlled epidural analgesia
  Arms: Study group
Device: Continuous infusion — Continuous infusion added to patient controlled epidural analgesia
  Arms: Control group

SUMMARY:
This study aims to establish if programmed intermittent epidural bolus combined to patient controlled analgesia in labour analgesia will lower the hourly bupivacaine consumption when compared to continuous infusion combined with patient controlled analgesia. The investigators' hypothesis is that the use of programmed intermittent epidural bolus will lower the hourly bupivacaine consumption.

DETAILED DESCRIPTION:
Patients are randomised to receive either a programmed bolus of 6ml each 45 minutes or a continuous infusion of 8ml/h. In each group, they have the possibility to add a PCEA bolus of 6ml every 20min as needed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant nulliparous or multiparous woman in labour
* Age ≥18 years
* Obtained consent for epidural analgesia
* ASA classification I-II-III
* Early labour (cervical dilation ≤6cm)

Exclusion Criteria:

* Pregnancy-related comorbidities (preeclampsia, eclampsia, gestational diabetes, large for gestational age fetus)
* Prematurity (<36 weeks of gestation)
* Multiple gestation
* Fentanyl allergy or hypersensitivity
* Patient unable to understand the PCEA
* Fetal breech position
* Maternal cardiac pathology and contraindication to Valsalva manoeuvre
* Patient with a pain visual analog scale (VAS) not ≤1/10 20 minutes after the anesthesiologist's initial bolus
* Intrathecal catheter or intravascular catheter
* Accidental dural puncture
* Patient refusal
* Patient with a history of chronic pain (pain lasting more than 3 months) or fibromyalgia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose of bupivacaine in milligrams per hour | 1 day
  Total dose of bupivacaine in milligrams divided by the total duration of the epidural in hours

SECONDARY OUTCOMES:
Evaluation of pain | 1 day
  Hourly pain measurement by visual analog scale, 0/10 being no pain and 10/10 being the worst pain imaginable
Anesthesiologist manual bolus | 1 day
  Total boluses by the anesthesiologist
PCEA boluses received | 1 day
  PCEA boluses received
PCEA boluses requested | 1 day
  PCEA boluses requested
Time lapse before the first PCEA request after the epidural connection | 1 day
  Time lapse before the first PCEA request after the epidural connection
First stage | 1 day
  Duration of the first stage of labour
Second stage | 1 day
  Duration of the second stage of labour
Assisted vaginal delivery | 1 day
  Number of assisted vaginal delivery (vacuum, forceps)
Cesarean section | 1 day
  Number of unplanned cesarean section
Motor blockade | 1 day
  Number of patients with a Bromage score ≥1
Patient satisfaction | 1 day
  Satisfaction of the analgesia provided by the epidural on a visual analog scale of 0-100, 0/100 being no satisfaction at all and 100/100 being entirely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Rivard, Dr., Principal Investigator — Université de Sherbrooke
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication for 5 years
Access Criteria: All access requests and criteria will be reviewed by the investigators of this study.

REFERENCES:
- [Background] Liu EH, Sia AT. Rates of caesarean section and instrumental vaginal delivery in nulliparous women after low concentration epidural infusions or opioid analgesia: systematic review. BMJ. 2004 Jun 12;328(7453):1410. doi: 10.1136/bmj.38097.590810.7C. Epub 2004 May 28. PMID 15169744
- [Background] Nunes J, Nunes S, Veiga M, Cortez M, Seifert I. A prospective, randomized, blinded-endpoint, controlled study - continuous epidural infusion versus programmed intermittent epidural bolus in labor analgesia. Braz J Anesthesiol. 2016 Sep-Oct;66(5):439-44. doi: 10.1016/j.bjane.2014.12.006. Epub 2015 Nov 19. PMID 27591455
- [Background] Salim R, Nachum Z, Moscovici R, Lavee M, Shalev E. Continuous compared with intermittent epidural infusion on progress of labor and patient satisfaction. Obstet Gynecol. 2005 Aug;106(2):301-6. doi: 10.1097/01.AOG.0000171109.53832.8d. PMID 16055579
- [Background] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Background] Lim Y, Sia AT, Ocampo C. Automated regular boluses for epidural analgesia: a comparison with continuous infusion. Int J Obstet Anesth. 2005 Oct;14(4):305-9. doi: 10.1016/j.ijoa.2005.05.004. PMID 16154735
- [Background] Lim Y, Chakravarty S, Ocampo CE, Sia AT. Comparison of automated intermittent low volume bolus with continuous infusion for labour epidural analgesia. Anaesth Intensive Care. 2010 Sep;38(5):894-9. doi: 10.1177/0310057X1003800514. PMID 20865875
- [Background] Fettes PD, Moore CS, Whiteside JB, McLeod GA, Wildsmith JA. Intermittent vs continuous administration of epidural ropivacaine with fentanyl for analgesia during labour. Br J Anaesth. 2006 Sep;97(3):359-64. doi: 10.1093/bja/ael157. Epub 2006 Jul 18. PMID 16849382
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Leo S, Ocampo CE, Lim Y, Sia AT. A randomized comparison of automated intermittent mandatory boluses with a basal infusion in combination with patient-controlled epidural analgesia for labor and delivery. Int J Obstet Anesth. 2010 Oct;19(4):357-64. doi: 10.1016/j.ijoa.2010.07.006. Epub 2010 Sep 15. PMID 20832282
- [Background] Tien M, Allen TK, Mauritz A, Habib AS. A retrospective comparison of programmed intermittent epidural bolus with continuous epidural infusion for maintenance of labor analgesia. Curr Med Res Opin. 2016 Aug;32(8):1435-40. doi: 10.1080/03007995.2016.1181619. Epub 2016 May 20. PMID 27100210
- [Background] Sia AT, Lim Y, Ocampo C. A comparison of a basal infusion with automated mandatory boluses in parturient-controlled epidural analgesia during labor. Anesth Analg. 2007 Mar;104(3):673-8. doi: 10.1213/01.ane.0000253236.89376.60. PMID 17312228
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] McKenzie CP, Cobb B, Riley ET, Carvalho B. Programmed intermittent epidural boluses for maintenance of labor analgesia: an impact study. Int J Obstet Anesth. 2016 May;26:32-8. doi: 10.1016/j.ijoa.2015.11.005. Epub 2015 Nov 27. PMID 26775896
- [Background] Epsztein Kanczuk M, Barrett NM, Arzola C, Downey K, Ye XY, Carvalho JC. Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Biased-Coin Up-and-Down Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 10 mL of Bupivacaine 0.0625% With Fentanyl 2 mug/mL. Anesth Analg. 2017 Feb;124(2):537-541. doi: 10.1213/ANE.0000000000001655. PMID 27755057
- [Background] Wong CA, McCarthy RJ, Hewlett B. The effect of manipulation of the programmed intermittent bolus time interval and injection volume on total drug use for labor epidural analgesia: a randomized controlled trial. Anesth Analg. 2011 Apr;112(4):904-11. doi: 10.1213/ANE.0b013e31820e7c2f. PMID 21430035
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Lee L, Dy J, Azzam H. Management of Spontaneous Labour at Term in Healthy Women. J Obstet Gynaecol Can. 2016 Sep;38(9):843-865. doi: 10.1016/j.jogc.2016.04.093. Epub 2016 Jun 25. PMID 27670710
- [Background] Todd KH, Funk JP. The minimum clinically important difference in physician-assigned visual analog pain scores. Acad Emerg Med. 1996 Feb;3(2):142-6. doi: 10.1111/j.1553-2712.1996.tb03402.x. PMID 8808375
- [Background] Singer AJ, Thode HC Jr. Determination of the minimal clinically significant difference on a patient visual analog satisfaction scale. Acad Emerg Med. 1998 Oct;5(10):1007-11. doi: 10.1111/j.1553-2712.1998.tb02781.x. PMID 9862594